CLINICAL TRIAL: NCT04719598
Title: Effects of Internet - Based Cognitive Behavioral Therapy on Sleep Quality Among a Sample of Saudi Postmenopausal Women
Brief Title: Effects of Internet - Based Cognitive Behavioral Therapy on Sleep Problems Among Sample of Post- Menopausal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Enas Mahrous AbdelAziz, Assistant professor, Jouf University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1384754968
Record Dates: First submitted 2020-12-25; First posted 2021-01-22 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Sleep Problem
Keywords: Post menopausal; intervention; sleep problems; CBT
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: one intervention group ( internet-based cognitive behavioral therapy) and one control group
Who Masked: Participant
Masking Description: all participants will randomly assign to either an internet-based group and control group through a generated computer selection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group is ( internet - based group) who will receive CBT sessions (Experimental): study group ( group A)
  Interventions: Behavioral: congnitive behavioural therapy
- control group ( group B) (No Intervention): researchers just answer their questions

INTERVENTIONS:
Behavioral: congnitive behavioural therapy — CBT Sessions divide into three main components; 1) cognitive interventions, concerns with cognitive restructuring attempts to change maladaptive thought about thoughts about sleep into more adaptable . 2) Behavioral intervention: concerns with Relaxation training, stimulus control, and sleep restriction promote relaxation and help to establish healthy sleep habits. 3) Psychoeducational interventions: Providing information about the connection between thoughts, feelings, behaviors, and sleep.
  Other Names: non
  Arms: intervention group is ( internet - based group) who will receive CBT sessions

SUMMARY:
Sleep problems become more prominent with aging and worse among post-menopause than perimenopause stage. The actual causes of sleep problems are unclear. However, it occurs commonly accompanied with or in the response of seriousness of menpausal symptoms as nocturnal hot flashes, mood disorders, and obstructive sleep apnea among menopauses. The Prevalence of sleep problems is variable ranged from 11.8 -62 % based on different studies.

Cognitive-behavioral therapy (CBT) is one of the short-term form of psychotherapy, used for managing sleep problems and insomnia , an efficacious as pharmacological treatment.

DETAILED DESCRIPTION:
As life expectancy has increased, women spend more than one-third of their lives in menopausal transition (MT) and the subsequent post menopause (PM).As a result of hormonal changes women experiences such symptoms as hot flashes, mood swings, anxiety, and sexual dysfunction that deteriorate their quality of life. Those symptoms usually begin in 45-53-year-olds and it varies in onset and severity from women to another and from country to another.

Symptoms of sleep problems include the difficulty of falling asleep, fractioned sleep, night-time awakening, the inability of resuming sleep, problems in waking up, fatigue, and daytime sleepiness that potentiate poor physical and mental quality of life.

The goal of CBT is to teach women how to modify maladaptive behaviors and thoughts that may contribute to a particular problem as sleep problems, anxious thoughts, and vasomotor symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Menopaused women age between 50 and65 years
2. Able to read and write
3. Being normally ( primary ) menopause at least one year
4. Willing to give written informed consent to participate in the study.
5. Women obtaining more than 5 of the total score of the Pittsburgh Sleep Quality Index (PSQI)( that indicates poor sleep )
6. Have smartphone with internet access (WhatsApp) application

Exclusion Criteria:

1. Has serious physical disorders or uncontrolled conditions as uncontrolled blood pressure , uncontrolled blood glucose level, on hemodialysis
2. Receiving psychotropic medications, hormone replacement therapy (HRT),
3. Undergoing hysterectomy
4. Has acute or chronic surgical conditions, cancer or any other serious illness
5. Has cognitive impairments or physical handicap
6. Giving prescribed or non-prescribed medication or herbals that influencing sleep .

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female post menpause ( 45-65 years)
Enrollment: 80 (Estimated)
Dates: Start 2021-01-25 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
change sleep quality post intervention | 8 weeks (two weeks ( introductory sessions ) pluse six weeks ( intervention sessions)
  improve quality of sleep than before intervention before intervention
change insomnia related to post menpausal symptoms post intervention | 8 weeks (two weeks ( introductory sessions ) pluse six weeks ( intervention sessions)
  decrease insomnia index score post intervention

SECONDARY OUTCOMES:
change menopausal symptoms post intervention | at the end of intervention program ( 8 weeks)
  decrease menopausal rating scale post intervention than pre intervention

IPD SHARING:
Plan to Share IPD: No